CLINICAL TRIAL: NCT05672108
Title: Phase II Trial of Lung Chemoemobolization
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22067; P30CA033572 (NIH); NCI-2022-10436 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22067 (Other: City of Hope Medical Center)
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Lung Non-Small Cell Carcinoma; Mediastinal Neoplasm; Pleural Neoplasm; Lung Metastases From Any Primary; Endobronchial Metastases; Colon Cancer; Sarcoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Mediastinal Neoplasms; Pleural Neoplasms; Colonic Neoplasms; Sarcoma | interventions — Ethiodized Oil; Iodized Oil; Mitomycin; Mitozytrex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Lung chemoembolization (Experimental): Patients receive lipiodol intra-arterially (IA), mitomycin IA, and embospheres IA and undergo TACE on study. Patients also undergo angiography and computed tomography (CT) at baseline and follow up.
  Interventions: Procedure: Computed Tomography; Drug: Ethiodized Oil; Drug: Mitomycin; Procedure: Transarterial Chemoembolization; Device: Tris-acryl Gelatin Microspheres

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Ethiodized Oil — Given IA
  Other Names: Ethiodol; Iodized Oil; Lipiodol
Drug: Mitomycin — Given IA
  Other Names: Ametycine; Jelmyto; MITO; Mito-C; Mito-Medac; Mitocin; Mitocin-C; Mitolem; Mitomycin C; Mitomycin-C; Mitomycin-X; Mitomycine C; Mitosol; Mitozytrex; Mutamycin; Mutamycine; NCI-C04706
Procedure: Transarterial Chemoembolization — Undergo TACE
  Other Names: TACE
Device: Tris-acryl Gelatin Microspheres — Given IA
  Other Names: Embospheres; TAGM; Trisacryl Gelatin Microspheres

SUMMARY:
This phase II trial evaluates how well transarterial chemoembolization (TACE) works for treating patients with non-small cell lung cancer or lung metastases. TACE is a minimally invasive procedure that involves injecting chemotherapy directly into an artery that supplies blood to tumors, and then blocking off the blood supply to the tumors. Mitomycin (chemotherapy), Lipiodol (drug carrier), and Embospheres (small plastic beads that block off the artery) are injected into the tumor-feeding artery. This traps the chemotherapy inside the tumor and also cuts off the tumor's blood supply. As a result, the tumor is exposed to a high dose of chemotherapy, and is also deprived of nutrients and oxygen. TACE can be effective at controlling or stopping the growth of lung tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine safety and efficacy (local progression free survival) of chemoembolization of lung cancer that is chemorefractory, unresectable, and unablatable.

OUTLINE:

Patients receive lung chemoembolization using Lipiodol, mitomycin, and Embospheres. Response to treatment is evaluated on computed tomography (CT) scans.

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer or lung metastases, with lung, endobronchial, pleural, or mediastinal tumors that are progressing on systemic therapy (or the patient cannot tolerate systemic therapy), and that are not amenable to resection, thermal ablation, or ablative radiation therapy
* Lung-dominant disease (majority of active tumor volume is in the chest)
* At least 18 years old

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status > 2
* Oxygen saturation < 92% on room air
* Forced expiratory volume in 1 second (FEV1) < 60%
* No measurable treatable disease, per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (for example, unable to measure tumor size on CT, or lung nodules are all < 1 cm)
* Life expectancy < 6 months
* Pulmonary hypertension (diagnosed or suspected on echocardiography, CT, magnetic resonance imaging [MRI], or direct pressure measurement)
* Recent pulmonary embolism (within 3 months)
* Pulmonary arteriovenous malformation
* Active lung infection (pneumonia, empyema, or lung abscess requiring therapy within 1 month)
* Symptomatic heart failure (American College of Cardiology [ACC]/American Heart Association [AHA] stage C or D)
* Left bundle branch block (contraindication to pulmonary angiography)
* Renal failure (estimated glomerular filtration rate [eGFR] < 30 mL/min/1.73 m^2)
* Pregnancy or intent to become pregnant
* Breast feeding
* Altered mental status that would interfere with consent or follow-up
* Platelets < 50,000 (after transfusion, if needed)
* International normalized ratio (INR) > 2 (after transfusion, if needed)
* Hemoglobin < 7 (after transfusion, if needed)
* Hyperthyroidism or history of hyperthyroidism, including subclinical hyperthyroidism (contraindication to lipiodol)
* Planned radioactive iodine imaging or therapy (contraindication to lipiodol)
* Allergy to lipiodol or mitomycin
* Allergy to iodinated contrast that cannot be treated with steroid / diphenhydramine premedication
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product, or that would affect subject safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2026-10-28 (Estimated); Study Completion 2026-10-28 (Estimated)

PRIMARY OUTCOMES:
Local progression free survival | Time from the initial transarterial chemoembolization (TACE) treatment to progression in a completely treated territory (or touching the border of a completely treated area), or death from any cause, assessed at 6 months
  Progression is determined using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. criteria, compared to the scan immediately prior to treatment of that territory, using the 2 largest measurable lesions per treated territory. Local progression-free survival will be estimated using the Kaplan-Meier method.
Incidence of adverse events | Up to 3 months after the last chemoembolization procedure
  Complications will be classified using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The rate of complications can be estimated with a standard error of less than 10%. Further, any complication that occurs with a 10% incidence will be observed with greater than 95% probability.

SECONDARY OUTCOMES:
Objective response rate (best response) | Within 3 months of treatment
  Evaluated on a per-treatment basis, using RECIST version 1.1 criteria.
Overall survival | Up to 9 months
  Will be estimated using the Kaplan-Meier method.
Progression-free survival | Up to 9 months
  Will be estimated using the Kaplan-Meier method.
Bronchial versus pulmonary artery blood supply | Up to 9 months
  Percentage of treatments where target tumors were supplied by bronchial artery, non-bronchial systemic artery, or pulmonary artery, based on catheter angiography. Confidence intervals of proportions will be estimated using the equal-tailed Jeffreys prior interval.
Lipiodol retention in treated tumors | 4-6 weeks post-procedure
  Correlation between lipiodol retention and change in tumor size will be evaluated using Spearman's rank correlation coefficient (rho) and Spearman's test.
Growth of TACE targeted lesions versus non-TACE targeted lesions | 4-6 weeks post-procedure
  Percentage change in size (largest diameter) of the largest treated, compared to the largest untreated tumor will be evaluated using the Wilcoxon signed-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Franz E Boas, MD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Boas FE, Salgia R, Waddington T, Massarelli E, Park JJ, Kessler J, Frankel P, Alexander ES, Solomon SB. Phase II Trial of Lung Chemoembolization. J Vasc Interv Radiol. 2023 Dec;34(12):2090-2092. doi: 10.1016/j.jvir.2023.08.006. Epub 2023 Aug 21. No abstract available. PMID 37611799